CLINICAL TRIAL: NCT05378334
Title: Efficacy and Safety of Bone-protecting and Mass-dispersesing Decoction (HuGuXiaoJiTang, HGXJT) Combining With ICIs in Bone Metastatic NSCLC Patients
Brief Title: Efficacy and Safety of HGXJT in Bone Metastatic NSCLC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Haibo Zhang, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021KT0613
Record Dates: First submitted 2022-04-04; First posted 2022-05-18 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Bone Metastatic; Immune Checkpoint Inhibitors; Chinese Formula; Efficacy; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Group (Experimental): Standard treatment: 4-6 cycles (3 weeks per cycle) of ICI + chemotherapy followed by ICI maintenance therapy, until tumor progression or at least 1 year.
  HGXJT decoction: 1 dose daily, until tumor progression or accumulation for 1 year.
  Interventions: Drug: ICI; Drug: Chemotherapy; Drug: Bone-protecting and Mass-dispersesing Decoction
- Control group (Placebo Comparator): Standard treatment: 4-6 cycles (3 weeks per cycle) of ICI + chemotherapy followed by ICI maintenance therapy, until tumor progression or at least 1 year.
  Placebo: 1 dose daily, until tumor progression or accumulation for 1 year.
  Interventions: Drug: ICI; Drug: Chemotherapy; Drug: Placebo

INTERVENTIONS:
Drug: ICI — PD-1 inhibitors selected by clinicians based on patients' condition
Drug: Chemotherapy — AP regimen（Pemetrexed 500mg/m2+carboplatin AUC=5,q3w） for non-squamous cancer patientsor or TP regimen（Paclitaxel 175mg/m2+carboplatin AUC=5, or albumin paclitaxel 100mg/m2+carboplatin AUC=5,q3w）for Squamous cancer patients.
Drug: Placebo — The particle size and color are similar to the HGXJT, and the smell and taste are close to the HGXJT, and the bacteria test is qualified
  Arms: Control group
Drug: Bone-protecting and Mass-dispersesing Decoction — Chinese Herbal Formula,also named as HGXJT
  Arms: Combination Group

SUMMARY:
This is a double-blind, randomized controlled study evaluating the efficacy and safety of HGXJT in combination with ICI-based standard treatment in lung cancer patients with bone metastases. Enrolled participates will randomly receive HGXJT or placebo during the first 4-6 cycles of ICI-based standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-small cell lung cancer diagnosed by histopathology or cytopathology.
2. Presence of bone metastases.
3. EGFR/ALK gene wild type.
4. No prior treatment with PD-1 inhibitors (combination or monotherapy)
5. Those who have not received prior antitumor therapy or have not received further antitumor therapy after failure of first-line antitumor therapy.
6. PS score (ECOG) ≤ 2 points
7. Normal hepatic and renal function.

   Normal hepatic function: total serum bilirubin level ≤ 1.5 times of the upper limit of normal value(ULN), serum serum aspartate aminotransferase(AST) & alanine aminotransferase(ALT) ≤ 2.5 times ULN

   Normal renal function: serum creatinine ≤ 1.5 mg/dl (133 μmol/L) and/or creatinine clearance ≥ 60 ml/min.
8. Presence of at least one assessable lesion.
9. Signed informed consent, patient willing to accept this regimen, able to adhere to the medication, and good compliance.

Exclusion Criteria:

1. Unable to complete the baseline assessment form
2. Combination of other serious illnesses, including uncontrolled active infection, severe electrolyte disturbances, and significant bleeding tendencies.
3. Pregnant or lactating women.
4. Combined autoimmune diseases, hematologic disorders, or long-term use of hormones or immunosuppressive drugs.
5. Combination of other uncontrolled tumors.
6. Combination of severe brain or mental illness that affects the patient's ability to self-report.
7. Combined organ transplant history (including bone marrow autotransplantation and peripheral stem cell transplantation).
8. Those who are legally incompetent and whose medical or ethical reasons affect the continuation of the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
(Disease control rate assessed by investigators) DCR (CR+PR+SD) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  DCR (disease control rate) is defined as sum of complete response (CR) rate, partial response (PR) rate and stable disease (SD) rate, according to RECIST v 1.1, based on the chest, abdomen and/or brain CT/MRI evaluation. Patients will undergo a follow-up imaging examination every 3 months, with an additional imaging examination after the first two cycles of treatment (normally 6 weeks).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  The time from the date of randomization to the date of disease progression, date of withdraw, or death from any cause, whichever occurs first.
Overall survival (OS) | From date of randomization to the date of withdraw or date of death from any cause, whichever occurs first, assessed up to 120 months.
  The time from the date of randomization to the date of withdraw or date of death from any cause, whichever occurs first.
ORR(Objective response rate) | From date of randomization until the date of death or date of withdraw, whichever came first, assessed up to 120 months
  ORR (overall response rate) is defined as sum of complete response (CR) rate and partial response (PR) rate , according to RECIST v 1.1, based on the chest, abdomen and/or brain CT/MRI evaluation. Patients will undergo a follow-up imaging examination every 3 months, with an additional imaging examination after the first two cycles of treatment (normally 6 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Professor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Proto C, Lo Russo G, Corrao G, Ganzinelli M, Facchinetti F, Minari R, Tiseo M, Garassino MC. Treatment in EGFR-mutated non-small cell lung cancer: how to block the receptor and overcome resistance mechanisms. Tumori. 2017 Jul 31;103(4):325-337. doi: 10.5301/tj.5000663. Epub 2017 Jul 1. PMID 28708233
- [Background] Zhong WZ, Zhou Q, Wu YL. The resistance mechanisms and treatment strategies for EGFR-mutant advanced non-small-cell lung cancer. Oncotarget. 2017 Aug 17;8(41):71358-71370. doi: 10.18632/oncotarget.20311. eCollection 2017 Sep 19. PMID 29050366
- [Background] Carbone DP, Reck M, Paz-Ares L, Creelan B, Horn L, Steins M, Felip E, van den Heuvel MM, Ciuleanu TE, Badin F, Ready N, Hiltermann TJN, Nair S, Juergens R, Peters S, Minenza E, Wrangle JM, Rodriguez-Abreu D, Borghaei H, Blumenschein GR Jr, Villaruz LC, Havel L, Krejci J, Corral Jaime J, Chang H, Geese WJ, Bhagavatheeswaran P, Chen AC, Socinski MA; CheckMate 026 Investigators. First-Line Nivolumab in Stage IV or Recurrent Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 22;376(25):2415-2426. doi: 10.1056/NEJMoa1613493. PMID 28636851
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Garon EB, Hellmann MD, Rizvi NA, Carcereny E, Leighl NB, Ahn MJ, Eder JP, Balmanoukian AS, Aggarwal C, Horn L, Patnaik A, Gubens M, Ramalingam SS, Felip E, Goldman JW, Scalzo C, Jensen E, Kush DA, Hui R. Five-Year Overall Survival for Patients With Advanced Non-Small-Cell Lung Cancer Treated With Pembrolizumab: Results From the Phase I KEYNOTE-001 Study. J Clin Oncol. 2019 Oct 1;37(28):2518-2527. doi: 10.1200/JCO.19.00934. Epub 2019 Jun 2. PMID 31154919
- [Background] Remon J, Passiglia F, Ahn MJ, Barlesi F, Forde PM, Garon EB, Gettinger S, Goldberg SB, Herbst RS, Horn L, Kubota K, Lu S, Mezquita L, Paz-Ares L, Popat S, Schalper KA, Skoulidis F, Reck M, Adjei AA, Scagliotti GV. Immune Checkpoint Inhibitors in Thoracic Malignancies: Review of the Existing Evidence by an IASLC Expert Panel and Recommendations. J Thorac Oncol. 2020 Jun;15(6):914-947. doi: 10.1016/j.jtho.2020.03.006. Epub 2020 Mar 14. PMID 32179179
- [Background] Chen Xian, Zhang Haibo, Liu Yihong, et al. Study on the correlation between the efficacy and NTX level of bone metastasis cancer pain treated with Bone Protecting and Anti-accumulation Formula combined with zoledronic acid and the evidence of kidney deficiency in Chinese medicine. New Chinese Medicine, 2017, 49(10): 117-120.
- [Background] Yang M, Lu J, Zhang G, Wang Y, He M, Xu Q, Xu C, Liu H. CXCL13 shapes immunoactive tumor microenvironment and enhances the efficacy of PD-1 checkpoint blockade in high-grade serous ovarian cancer. J Immunother Cancer. 2021 Jan;9(1):e001136. doi: 10.1136/jitc-2020-001136. PMID 33452206
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Drilon A, Wolchok JD, Carvajal RD, McHenry MB, Hosein F, Harbison CT, Grosso JF, Sznol M. Five-Year Survival and Correlates Among Patients With Advanced Melanoma, Renal Cell Carcinoma, or Non-Small Cell Lung Cancer Treated With Nivolumab. JAMA Oncol. 2019 Oct 1;5(10):1411-1420. doi: 10.1001/jamaoncol.2019.2187. PMID 31343665
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Ferrara R, Mezquita L, Texier M, Lahmar J, Audigier-Valette C, Tessonnier L, Mazieres J, Zalcman G, Brosseau S, Le Moulec S, Leroy L, Duchemann B, Lefebvre C, Veillon R, Westeel V, Koscielny S, Champiat S, Ferte C, Planchard D, Remon J, Boucher ME, Gazzah A, Adam J, Bria E, Tortora G, Soria JC, Besse B, Caramella C. Hyperprogressive Disease in Patients With Advanced Non-Small Cell Lung Cancer Treated With PD-1/PD-L1 Inhibitors or With Single-Agent Chemotherapy. JAMA Oncol. 2018 Nov 1;4(11):1543-1552. doi: 10.1001/jamaoncol.2018.3676. PMID 30193240
- [Background] Ferrara R, Mezquita L, Texier M, et al. Fast-progression(FP), hyper-progression(HPD) and early deaths(ED) in advanced non-small cell lung cancer (NSCLC) patients(pts) upon PD-(L)-1 blockade (IO). J Clin Oncol, 2019, 37(suppl 15), 9107.
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Wu YL, Lu S, Cheng Y, Zhou C, Wang J, Mok T, Zhang L, Tu HY, Wu L, Feng J, Zhang Y, Luft AV, Zhou J, Ma Z, Lu Y, Hu C, Shi Y, Baudelet C, Cai J, Chang J. Nivolumab Versus Docetaxel in a Predominantly Chinese Patient Population With Previously Treated Advanced NSCLC: CheckMate 078 Randomized Phase III Clinical Trial. J Thorac Oncol. 2019 May;14(5):867-875. doi: 10.1016/j.jtho.2019.01.006. Epub 2019 Jan 17. PMID 30659987
- [Background] Vokes EE, Ready N, Felip E, Horn L, Burgio MA, Antonia SJ, Aren Frontera O, Gettinger S, Holgado E, Spigel D, Waterhouse D, Domine M, Garassino M, Chow LQM, Blumenschein G Jr, Barlesi F, Coudert B, Gainor J, Arrieta O, Brahmer J, Butts C, Steins M, Geese WJ, Li A, Healey D, Crino L. Nivolumab versus docetaxel in previously treated advanced non-small-cell lung cancer (CheckMate 017 and CheckMate 057): 3-year update and outcomes in patients with liver metastases. Ann Oncol. 2018 Apr 1;29(4):959-965. doi: 10.1093/annonc/mdy041. PMID 29408986
- [Background] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Vandormael K, Riccio A, Yang J, Pietanza MC, Brahmer JR. Updated Analysis of KEYNOTE-024: Pembrolizumab Versus Platinum-Based Chemotherapy for Advanced Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score of 50% or Greater. J Clin Oncol. 2019 Mar 1;37(7):537-546. doi: 10.1200/JCO.18.00149. Epub 2019 Jan 8. PMID 30620668
- [Background] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- [Background] Hellmann MD, Ciuleanu TE, Pluzanski A, Lee JS, Otterson GA, Audigier-Valette C, Minenza E, Linardou H, Burgers S, Salman P, Borghaei H, Ramalingam SS, Brahmer J, Reck M, O'Byrne KJ, Geese WJ, Green G, Chang H, Szustakowski J, Bhagavatheeswaran P, Healey D, Fu Y, Nathan F, Paz-Ares L. Nivolumab plus Ipilimumab in Lung Cancer with a High Tumor Mutational Burden. N Engl J Med. 2018 May 31;378(22):2093-2104. doi: 10.1056/NEJMoa1801946. Epub 2018 Apr 16. PMID 29658845
- [Background] Hellmann MD, Paz-Ares L, Bernabe Caro R, Zurawski B, Kim SW, Carcereny Costa E, Park K, Alexandru A, Lupinacci L, de la Mora Jimenez E, Sakai H, Albert I, Vergnenegre A, Peters S, Syrigos K, Barlesi F, Reck M, Borghaei H, Brahmer JR, O'Byrne KJ, Geese WJ, Bhagavatheeswaran P, Rabindran SK, Kasinathan RS, Nathan FE, Ramalingam SS. Nivolumab plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2019 Nov 21;381(21):2020-2031. doi: 10.1056/NEJMoa1910231. Epub 2019 Sep 28. PMID 31562796
- [Background] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Background] Gadgeel S, Rodriguez-Abreu D, Speranza G, Esteban E, Felip E, Domine M, Hui R, Hochmair MJ, Clingan P, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Garon EB, Novello S, Rubio-Viqueira B, Boyer M, Kurata T, Gray JE, Yang J, Bas T, Pietanza MC, Garassino MC. Updated Analysis From KEYNOTE-189: Pembrolizumab or Placebo Plus Pemetrexed and Platinum for Previously Untreated Metastatic Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2020 May 10;38(14):1505-1517. doi: 10.1200/JCO.19.03136. Epub 2020 Mar 9. PMID 32150489
- [Background] Jenkins RW, Thummalapalli R, Carter J, Canadas I, Barbie DA. Molecular and Genomic Determinants of Response to Immune Checkpoint Inhibition in Cancer. Annu Rev Med. 2018 Jan 29;69:333-347. doi: 10.1146/annurev-med-060116-022926. Epub 2017 Nov 3. PMID 29099676
- [Background] Wellenstein MD, de Visser KE. Cancer-Cell-Intrinsic Mechanisms Shaping the Tumor Immune Landscape. Immunity. 2018 Mar 20;48(3):399-416. doi: 10.1016/j.immuni.2018.03.004. PMID 29562192
- [Background] Stankovic B, Bjorhovde HAK, Skarshaug R, Aamodt H, Frafjord A, Muller E, Hammarstrom C, Beraki K, Baekkevold ES, Woldbaek PR, Helland A, Brustugun OT, Oynebraten I, Corthay A. Immune Cell Composition in Human Non-small Cell Lung Cancer. Front Immunol. 2019 Feb 1;9:3101. doi: 10.3389/fimmu.2018.03101. eCollection 2018. PMID 30774636
- [Background] Bremnes RM, Busund LT, Kilvaer TL, Andersen S, Richardsen E, Paulsen EE, Hald S, Khanehkenari MR, Cooper WA, Kao SC, Donnem T. The Role of Tumor-Infiltrating Lymphocytes in Development, Progression, and Prognosis of Non-Small Cell Lung Cancer. J Thorac Oncol. 2016 Jun;11(6):789-800. doi: 10.1016/j.jtho.2016.01.015. Epub 2016 Feb 1. PMID 26845192
- [Background] Chaft JE, Hellmann MD, Velez MJ, Travis WD, Rusch VW. Initial Experience With Lung Cancer Resection After Treatment With T-Cell Checkpoint Inhibitors. Ann Thorac Surg. 2017 Sep;104(3):e217-e218. doi: 10.1016/j.athoracsur.2017.03.038. PMID 28838509
- [Background] Gettinger SN, Wurtz A, Goldberg SB, Rimm D, Schalper K, Kaech S, Kavathas P, Chiang A, Lilenbaum R, Zelterman D, Politi K, Herbst RS. Clinical Features and Management of Acquired Resistance to PD-1 Axis Inhibitors in 26 Patients With Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2018 Jun;13(6):831-839. doi: 10.1016/j.jtho.2018.03.008. Epub 2018 Mar 22. PMID 29578107
- [Background] Turpin A, Duterque-Coquillaud M, Vieillard MH. Bone Metastasis: Current State of Play. Transl Oncol. 2020 Feb;13(2):308-320. doi: 10.1016/j.tranon.2019.10.012. Epub 2019 Dec 23. PMID 31877463
- [Background] Limones A, Saez-Alcaide LM, Diaz-Parreno SA, Helm A, Bornstein MM, Molinero-Mourelle P. Medication-related osteonecrosis of the jaws (MRONJ) in cancer patients treated with denosumab VS. zoledronic acid: A systematic review and meta-analysis. Med Oral Patol Oral Cir Bucal. 2020 May 1;25(3):e326-e336. doi: 10.4317/medoral.23324. PMID 32271321
- [Background] Xiang L, Gilkes DM. The Contribution of the Immune System in Bone Metastasis Pathogenesis. Int J Mol Sci. 2019 Feb 25;20(4):999. doi: 10.3390/ijms20040999. PMID 30823602
- [Background] Jiao S, Subudhi SK, Aparicio A, Ge Z, Guan B, Miura Y, Sharma P. Differences in Tumor Microenvironment Dictate T Helper Lineage Polarization and Response to Immune Checkpoint Therapy. Cell. 2019 Nov 14;179(5):1177-1190.e13. doi: 10.1016/j.cell.2019.10.029. PMID 31730856
- [Background] Owen KL, Parker BS. Beyond the vicious cycle: The role of innate osteoimmunity, automimicry and tumor-inherent changes in dictating bone metastasis. Mol Immunol. 2019 Jun;110:57-68. doi: 10.1016/j.molimm.2017.11.023. Epub 2017 Nov 27. PMID 29191489
- [Background] Chen Yunying,Wu Danhong. Combination of Chinese and Western medicine in the treatment of painful bone metastases in 3O cases. Fujian Traditional Chinese Medicine, 2001, 32:1.
- [Background] Niu Wei, Wu Wangen. Advances in Chinese medicine treatment of bone metastatic cancer. Chinese Medicine Research, 2001,14:53.
- [Background] Cui Yiwen, Wang Jie, Chen Teng. Research progress of Chinese medicine in regulating tumor immune response. Tumor, 2019, 39, 674-679.